CLINICAL TRIAL: NCT02115685
Title: Sympathetic-Somatomotor Coupling in Human Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: Marquette University (Other)
Responsible Party: Principal Investigator, Thomas G Hornby, PT, PhD, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01NS079751 (NIH)
Record Dates: First submitted 2014-04-14; First posted 2014-04-16 (Estimated); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: Spinal Cord Injury
Keywords: spinal cord injury; sympathetic nervous system; locomotor training; exercise
MeSH Terms: conditions — Spinal Cord Injuries; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- One day testing (No Intervention): Aim 1 will be to measure bloodflow during exercise of the legs (below the injury). This aim will examine the control of bloodflow and muscle contractions and how it changes after spinal cord injury.
- Effects of long term training (Experimental): Aim 3 will then look at changes in bloodflow during exercise after training. Three different eight week exercise training programs will be tested including 1) treadmill training at high intensity as defined by 70-80% of HRR or 15-17 RPE 2) treadmill training at low intensity as defined by 30-40% of HRR or <13 RPE
  Interventions: Other: Treadmill Training

INTERVENTIONS:
Other: Treadmill Training — Subjects will be randomized to a high intensity and low intensity group. The high intensity group will train at 70-80% of their HRR and the low intensity group will train at 30-40% of their HRR.
  Arms: Effects of long term training

SUMMARY:
Significance: The long term objective of this study is to improve physical therapy and fitness programs in people with spinal cord injury. The results of the study will demonstrate the importance of matching blood flow to a muscle with exercise of that same muscle.

Scientific Objective: The objective of the study is to measure how the body regulates bloodflow to a muscle during exercise. We intend to study these effects by triggering blood flow changes during movement, and measuring bloodflow changes during exercise in people with spinal cord injury. We will also look at the long term effects of different exercise programs on bloodflow during exercise.

Study Populations: This study will involve people with partial spinal cord injury and age and sex matched controls without injury.

Specific Aims: Aim 1 will be to measure bloodflow during exercise of the legs (below the injury). This aim will examine the control of bloodflow and muscle contractions and how it changes after spinal cord injury. Aim 2 will then look at changes in bloodflow during exercise after training. Three different eight week exercise training programs will be tested including 1) upper body ergometry, 2) treadmill training with exertion level matched to the upper body ergometry and 3) treadmill training with heart rate matched to an initial test of upper body ergometry.

DETAILED DESCRIPTION:
The regulation of cardiovascular systems during muscle activity is poorly understood in people with incomplete spinal cord injury (SCI). In the past, disruptions in somatomotor and sympathetic control have been investigated separately in SCI. We propose to investigate the coupling of sympathetic and somatomotor control because it is relevant to exercise training paradigms that are designed to improve somatomotor function or enhance physical fitness. Our approach will be to measure tendon tap reflexes, voluntary muscle activation, and blood flow of the knee (below injury) and elbow (above injury) before and after sympathetic stimuli consisting of cold pressor tests, mental math and an acute bout of exercise. These data will provide information about sympathetic control of blood flow during muscle activity. Plasticity of the sympatheticsomatomotor coupling will also be investigated by making measurements before and after a treadmill training exercise program. These experiments will enable us to address three aims. Aim 1 will be to characterize coupling of sympathetic and somatomotor systems below the level of spinal injury. This aim will examine spinal sympathetic and motor reflexes and their interactions. It will also examine how descending somatomotor coupling is disrupted by the spinal injury. In Aim 2, we will identify changes in the interactions of sympathetic and somatomotor systems above a spinal injury. Because of the injury and the changes that occur below the injury, the sympathetic-somatomotor coupling is also likely to be disrupted in the arm. Aim 3 will then demonstrate plasticity of sympathetic-somatomotor coupling after exercise training. Three different eight week exercise training programs will be tested including 1) treadmill training with exertion level matched to 70-80% of HRR 2)treadmill training with 30-40% HRR. The exercise training will be tested in a randomized crossover study design with one month between exercise training paradigms. We anticipate that there will be plasticity of sympathetic-somatomotor coupling and that the exercise training effects will normalize control of these systems. However, because of the injury, we anticipate that adaptations will differ from non-injured controls.

This study has implications for exercise training in human SCI. The coupling of sympathetic and somatomotor systems is expected to depend on whether exercise targets the upper or lower body. The recovery of function requires both the improvement in the control of movement as well as in the regulation of blood flow to active muscle groups. In addition, this study is important for understanding the potential impact of treadmill exercise training on cardiovascular fitness, a topic of increasing interest in people with limitations to physical activity.

ELIGIBILITY:
Inclusion Criteria:

* incomplete SCI
* subjects will be over age 18
* to fit in the apparatus and to assure a mature gait pattern
* at least 6 months post injury, and medically stable with an incomplete lesion between levels T1-T10
* lower extremity motor score of 10 or greater
* presence of intact stretch reflexes, detected clinically
* no previous history or evidence of peripheral nerve damage in the lower extremities
* Subjects must be able to step on a treadmill with no more than 40% body weight support.

Healthy controls will be age and sex matched to the subjects with spinal cord injury.

Exclusion Criteria:

* unhealed decubiti,
* bladder or other infection
* severe contracture or osteoporosis
* heterotopic ossification
* cardiac arrhythmia
* inability to give informed consent
* an episode of autonomic dysreflexia in the past year
* use of spasticity or cardiovascular medications (e.g. baclofen)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-04; Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Arterial blood flow | 6 hours
  Subject will be tested with doppler ultrasonography immediately pre and post sympathetic stressor. Testing sessions will take anywhere between 3-6 hours.

SECONDARY OUTCOMES:
Graded Treadmill Exercise Test | 15 months
  Graded treadmill exercise test will be tested at multiple intervals pre and post training paradigms.
Heart rate | 15 months
  Heart rate will be tested continuously during sympathetic stressors and at multiple intervals pre and post training paradigms with a Finapres.
Knee torque | 8 hours
  Knee torque will be tested with the Biodex both pre and post sympathetic stressors.
Tendon tap reflexes | 8 hours
  Tendon tap reflexes will be tested during one day testing pre and post sympathetic stressors.

CONTACTS AND LOCATIONS:
Overall Officials: Brian D Schmidt, MD, Principal Investigator — Marquette University; George Hornby, PT, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- Rehabilitation Institute of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Lotter JK, Henderson CE, Plawecki A, Holthus ME, Lucas EH, Ardestani MM, Schmit BD, Hornby TG. Task-Specific Versus Impairment-Based Training on Locomotor Performance in Individuals With Chronic Spinal Cord Injury: A Randomized Crossover Study. Neurorehabil Neural Repair. 2020 Jul;34(7):627-639. doi: 10.1177/1545968320927384. Epub 2020 Jun 1. PMID 32476619